CLINICAL TRIAL: NCT05133063
Title: The Impact of a Gratitude Intervention on Stress Reactivity: A Randomised Control Trial
Brief Title: The Impact of a Gratitude Intervention on Stress Reactivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Maynooth (Other)
Collaborators: Bial Foundation (Unknown); Dr. Brenda O'Connell (Unknown); Dr. Deirdre O'Shea (Unknown)
Responsible Party: Principal Investigator, Brian Leavy, Principle Investigator, National University of Ireland, Maynooth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20501892
Record Dates: First submitted 2021-10-05; First posted 2021-11-24 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Positive Emotions; Blood Pressure; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude intervention (Experimental): Participants will complete a gratitude letter where they spend eight minutes writing a letter of gratitude. The individual writes about his feelings of gratitude through a letter, based on a written instruction.
  Interventions: Behavioral: Gratitude letter
- Control intervention. (Active Comparator): Participants spend eight minutes writing a note describing the lab in which the study is being run.
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: Gratitude letter — Participants are given the following instructions:
  Think of someone in your life who you feel like you have never fully or properly thanked for something meaningful or important that they did for you. . . . In the space provided below, please write a note to this person that describes why you feel like you never properly thanked them and letting them know why you feel thankful for something important that they did for you. Though this letter will not actually be sent to this person and is simply an exercise for you, please use this as an opportunity to really explore those feelings surrounding how you feel about what they have done for you and write honestly and openly from your heart. You have ten minutes.
  Arms: Gratitude intervention
Behavioral: Control intervention — Participants receive the following instructions:
  Think of the room you are in…. In the space below, please provide a description of the room you are in. Try to focus on the specific elements in the room, the colours of the wall or objects in the room. Use this writing session as an opportunity to paint a detailed picture of this room and include as much specific information as you can. You have ten minutes.
  Arms: Control intervention.

SUMMARY:
This study will employ a randomized mixed between-within experimental stress-testing protocol design. Physiological responses (blood pressure and pulse) will be recorded throughout a baseline, gratitude induction, standard stress-task and recovery period. Participants will be randomly allocated to the experimental (grateful induction) or control condition (neutral induction). Gratitude will be induced by completing a gratitude letter. Demographics will be measured. Psychosocial and health variables will be measured psychometrically at baseline to assess pre-existing levels and after both manipulations (allocated induction and stress task) to monitor expected change over time between conditions. Stress task is an adapted version of the Trier Stress Testing protocol.

DETAILED DESCRIPTION:
This study will employ an experimental within-subjects design, in which all participants are exposed to the same task and measures. The study will take place in Cubicle 1 of the Psychology Department, 2nd floor John Hume Building. On entry into the lab, participants will first be required to read the study information sheet and provide informed consent before the formal testing session begins. This standard protocol will comprise of the collection of demographic information, the administration of questionnaires (See supporting documentation) and the monitoring of physiological responses. The monitoring phase involves the following periods, a 20 minute acclimatisation, 10 minute baseline, 8 minute intervention, a 12-stress task and a 10 minute recovery period. During baseline general socio-demographic and lifestyle information will be collected through standard questionnaires (e.g. age, gender, height smoking status, health status and family history pertaining to the cardiovascular system; see supporting documentation). If predictive of blood pressure in the current study all potential confounds will be controlled for statistically in relevant analyses to isolate the contribution of the predictor variables, in this case state and trait gratitude, to the cardiovascular changes. Physiological responses -systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR)- will be measured noninvasively using a GE Dinamap Pro 400 and will be recorded throughout with a standard blood pressure cuff placed over the brachial artery on the participant's non-dominant arm. During the baseline phase psychological variables will be measured psychometrically.

Following this baseline phase, participants will randomly be allocated to either the control or experimental condition. The experimental condition will involve writing a letter thanking someone the participant had not thanked before. The control group will complete a writing exercise wherein they describe the laboratory room. They will have 8 minutes to complete this.

Following this intervention phase, participants will then complete an adapted form of the widely used Trier Social Stress Test, which involves participants subtracting numbers out loud and giving a short speech wherein they describe three of their best and worst characteristics . After the stress task, in the recovery phase participants will answer a series of questions pertaining to how they found the stress task. They will then sit for 8 minutes while recovery measures are taken.

Following this, all participants will be fully debriefed (supporting documentation) and thanked for their participation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to consent

Exclusion Criteria:

* Participants with a diagnosis of cardiovascular disease, hypertension, oran immune disorder
* Participants who are pregnant.
* Participants taking medication inﬂuencing cardiovascular measures.
* Participants who consumed alcohol 12 hours before study.
* Participants who exercised 12 hours before study.
* Participants who consumed nicotine 2 hours before study.
* Participants who consumed caffeine 2 hours before study.
* Participants who ate 1 hour before study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood pressure reactivity | Measured over the course of the study (1 hour)
  This will be done by taking the mean of the baseline measures and subtracting it from the mean of the stress task measures.
Diastolic Blood pressure reactivity | Measured over the course of the study (1 hour)
  This will be done by taking the mean of the baseline measures and subtracting it from the mean of the stress task measures.
Heart rate reactivity | Measured over the course of the study (1 hour)
  This will be done by taking the mean of the baseline measures and subtracting it from the mean of the stress task measures.
Systolic Recovery | Measured over the course of the study (1 hour)
  This will be done by taking the mean of the baseline measures and subtracting it from the mean of the recovery measures taken after the stress task.
Diastolic Recovery | Measured over the course of the study (1 hour)
  This will be done by taking the mean of the baseline measures and subtracting it from the mean of the recovery measures taken after the stress task.
Heart Rate Recovery | Measured over the course of the study (1 hour)
  This will be done by taking the mean of the baseline measures and subtracting it from the mean of the recovery measures taken after the stress task.

CONTACTS AND LOCATIONS:
Locations (1):
- Maynooth Univeristy, Maynooth, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No